CLINICAL TRIAL: NCT04042805
Title: Sintilimab Combined With Lenvatinib in Local Advanced Hepatocellular Carcinoma: A Single-arm, Open-label, Phase II Clinical Study
Brief Title: Sintilimab Combined With Lenvatinib in Local Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baocai Xing (Other)
Responsible Party: Sponsor-Investigator, Baocai Xing, Professor, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019088
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab Plus Lenvatinib (Experimental): Participants receive lenvatinib 12 mg (for participants with screening body weight ≥60 kg) or 8 mg (for participants with screening body weight <60 kg) orally once a day (QD) plus sintilimab 200 mg intravenously every 3 weeks up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Interventions: Biological: Sintilimab; Drug: Lenvatinib

INTERVENTIONS:
Biological: Sintilimab — 200mg intravenously every 3 weeks
  Other Names: IBI308
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing.

SUMMARY:
This ia a single-arm, single-center, not-randomized, open-label phase II study. The purpose of this study is to evaluate the efficacy and safety of Sintilimab (PD-1 antibody) combined with Lenvatinib(TKI) for the treatment of local advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of hepatocellular carcinoma confirmed by radiology, histology, or cytology
* Barcelona Clinic Liver Cancer (BCLC) Stage C disease without any distant or lymphatic metastasis , or BCLC Stage B disease not amenable to curative surgery
* No previous systemic anticancer treatment or TACE treatment
* Age ≥18 years
* ECOG performance status: 0-1
* Child Pugh score≤7
* Has at least one measurable hepatocellular carcinoma (HCC) lesion based on RECIST 1.1
* Life expectancy ≥12 weeks.
* Patients must be able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Fibrous lamina hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma
* History of hepatic encephalopathy or liver transplantation
* Pleural effusion, ascites and pericardial effusion with clinical symptoms or needing drainage.
* Untreated hepatitis infection: HBV DNA>2000IU/mlor10000 copy/ml, HCV RNA> 1000copy/ml, both HbsAg and anti-HCV body are positive.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* History of symptomatic interstitial lung disease or other conditions that may cause confusion when discovering or managing suspicious drug-related lung toxicity
* With serious systemic diseases such as heart disease and cerebrovascular disease, and the condition is unstable or uncontrollable.
* Evidence of active pulmonary tuberculosis (TB).
* Positive test of immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)
* History of allergic reactions to related drugs
* Pregnant women, nursing mothers

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 1 year after the last patient's enrollment

SECONDARY OUTCOMES:
Overall Survival | 2 years after the last patient's enrollment
Safety of combination sintilimab and lenvatinib as evaluated by incidence of adverse events(AEs), serious adverse events (SAEs). | 2 years after the last patient's enrollment
Conversion rate to surgery | 1 year after the last patient's enrollment
  Conversion rate defined as the proportion of participants be able to receive surgery after the initiation of the study treatment
Tumor mutation burden in association with ORR and survival. | 1 year after the last patient's enrollment
  It will be performed by NGS.

CONTACTS AND LOCATIONS:
Overall Officials: Baocai Xing, Doctor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China